CLINICAL TRIAL: NCT05226208
Title: Predictors of Severe Labor Pain: Prospective Observational Study
Brief Title: Labour Pain is a Subjective Experience. The Degree of a Woman's Suffering in Childbirth Depends on Indirect Factors
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Anastasiia Romanenko, MD, Principal Investigator, Bogomolets National Medical University
Other Study IDs: 0002-9033-149X
Record Dates: First submitted 2021-11-20; First posted 2022-02-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pain, Labor
Keywords: labor pain; antenatal education; support by doula
MeSH Terms: conditions — Labor Pain | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with not severe labour pain: Group 1 included 282 patients (pain level ≥7 mm according to the VAS).
  Interventions: Diagnostic Test: Visual analogue scale (VAS); Diagnostic Test: General anxiety scale (GAD-2) and survey
- Women with severe labour pain: Group 2 included 84 patients (pain level ≤ 6 mm using the VAS).
  Interventions: Diagnostic Test: Visual analogue scale (VAS); Diagnostic Test: General anxiety scale (GAD-2) and survey

INTERVENTIONS:
Diagnostic Test: Visual analogue scale (VAS) — In the postpartum period all patients filled VAS and underwent interviews from the 1st to the 3rd day after delivery.
Diagnostic Test: General anxiety scale (GAD-2) and survey — In the postpartum period all patients filled survey with GAD-2 and underwent interviews from the 1st to the 3rd day after delivery.

SUMMARY:
Pain During Childbirth is a Complex and Subjective Experience. The Degree of a Woman's Suffering in Childbirth Depends on the Intensity of Labour Pain and Many Indirect Factors. Complex Interrelated Effects on Labour Pain Are Limited by the Little Number of Studies Available. That is Why it is Necessary to Determine the Probable Factors That May Affect the Intensity of Pain.

DETAILED DESCRIPTION:
A prospective observational study was conducted in the period from December 2020 to May 2021 at the Kyiv City Maternity Hospital №5 (Kyiv, Ukraine). The study protocol was approved by the Bogomolets National Medical University Ethics Committee. The examined predictors were derived from mothers' self-report of overall childbirth. 366 women took part in research, 282 of participants rated their pain by ≤ 60 mm visual analog scale (VAS), while 84 patients reported their pain by ≥70 mm VAS. The aim of study was to investigate predictors of severe labour pain. In the postpartum period all patients filled questionnaires and underwent interviews from the 1st to the 3rd day after delivery. The following groups of risk factors were studied:

1. Demographic indicators (age, level of working capacity 2 months before childbirth, attendance of maternity school).
2. General level of health (woman's level of health before childbirth, daily physical activity before childbirth, bad habits - smoking during pregnancy).
3. Presence of mental disorders before childbirth (level of anxiety 2 weeks before childbirth, widespread muscle pain with fatigue or problems with memory, sleep, and mood).
4. The presence of chronic pain, chronic headache or chronic back pain, the presence of rheumatoid arthritis during pregnancy, the presence of increased intracranial pressure during pregnancy.
5. Presence of chronic intestinal diseases (irritable bowel syndrome).
6. The level of assistance during childbirth (constant support of the doula during childbirth, the woman's ability to control pain in childbirth).

ELIGIBILITY:
Inclusion Criteria:

* mothers over 18 years of age, 1st or 2nd parturitions, childbirth with the birth of the alive fetus.

Exclusion Criteria:

* mothers over 45 years of age, inability to obtain the informed consent of the patient or his legal representative.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — mothers over 18 years of age
Study Population: mothers over 18 years of age, 1st or 2nd parturitions, childbirth with the birth of the alive fetus
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Prenatal anxiety level | 6 months
  Generalized Anxiety Disorder-2 scale is a tool, which confirms the diagnosis of generalized anxiety disorder. A positive Generalized Anxiety Disorder-2 scale result is a score of at least 3 points. It is considered to be negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, PhD, Study Director — Bogomolets National Medical University; Dmytro Govsieiev, PhD, Study Director — Bogomolets National Medical University; Kateryna Bielka, PhD, Study Chair — Bogomolets National Medical University; Anastasiia Romanenko, MD, Principal Investigator — Bogomolets National Medical University
Locations (1):
- Bogomolets National Medical University, Kiev, Ukraine

REFERENCES:
- See also: World Health Organization (WHO). Intrapartum care for a positive childbirth experience: a practical guide. Accessed 7 February 2018. — https://www.who.int/publications/i/item/9789241550215